## **Treatment during pregnancy Consent Form**

Version 4.3 Version Date: 05 Jul 2022 SUBJECT IDENTIFICATION

Protocol Title: endTB-Q (Evaluating Newly Approved Drugs in Combination Regimens for

Multidrug-Resistant TB with Fluoroquinolone Resistance)

Sponsor: Médecins Sans Frontières (Doctors Without Borders) – France

Principal Investigators: Carole Mitnick, Sc.D. and Lorenzo Guglielmetti, M.D.

Site Principal Investigator: [Insert PI Name]
Research Center: [Insert Research Center Name]

| Participant Name (please print): |
|----------------------------------|
| Study Subject ID: |

#### About this consent form

We are asking you to read this form because you are currently receiving study drugs to treat your tuberculosis ("TB") as part of the endTB-Q clinical trial, you are at least 18 years of age, and because you are now pregnant. Please read this form carefully. The purpose of this form is to request your consent to continue participating in the study. A member of the study team will also explain to you verbally the information provided in this form.

When you initially consented to participate into the study, we explained that we don't know if some of the study drugs given in the study are safe if taken during pregnancy. We explained that pregnant women cannot enter the study and we asked you to use birth control while taking the study drugs.

After the \_\_\_\_\_ dose of the study treatment \_\_\_\_\_, but before treatment was complete, we learned that you are pregnant. Your study doctor believes that there are more benefits than risks for you to stay in the study. Since your condition has changed, we are asking again if you are still willing to participate in the study.

If you have any questions about the information provided, about the reason we are asking for your consent or about this form, please ask us. Signing this form is voluntary; it is up to you to decide whether you will stay in the study and keep receiving the study drugs without terminating the pregnancy. If you agree, we will ask you to sign this form to confirm that you want to continue. We will give you a signed copy of this form to keep. You can decide to stop taking part in this study at any time if you do not want to, even after signing this form.

If you are not able to sign the consent form, but you would like to participate, you can ask someone you know to sign for you and you can make a thumbprint to show that you understand and would like to continue taking part.

#### Why is it proposed that I stay in the study even though I'm pregnant?

The effects of your study treatment on pregnancy and on the developing fetus (baby still in the womb) are currently not known or not fully understood.

However, based on the information now available about your clinical condition, the drugs you are taking, and your treatment options if you choose to leave the study, your study doctor believes that the expected benefits of continuing to receive the study drugs are bigger than the risks for you and your baby.

#### Will I be told why the doctor thinks I should stay in the study?

Based on the TB study drugs you are currently taking and your clinical condition, your study doctor will explain you why s/he has proposed that you stay in the study.

# **Treatment during pregnancy Consent Form**

Version 4.3 Version Date: 05 Jul 2022

SUBJECT IDENTIFICATION

In detail s/he will explain all the options available to you:

- o the available information about the safety of taking these drugs during pregnancy;
- o the possible risks and benefits to you and your baby if you stay in the study;
- o the possible risks and benefits to you and your baby if you leave the study;
- o the possible (treatment) options you might have if you leave the study; and
- o the possible risks to you and your baby from your TB disease if you decide to stop taking TB treatment completely.

If the explanation is not clear, we want you to ask questions until everything is clear and you have sufficient information and time to take your decision.

#### What will happen during the study, if I decide to remain in the study?

You will be monitored using the same schedule you agreed to when you signed the original research consent form for endTB-Q clinical trial.

If you decide to stay in the study, your study doctor will talk to you, and, if you permit, your gynaecologist and/or obstetrician (doctor in charge of pregnant women), to make sure the development of your baby is closely followed during the whole pregnancy.

We would also like to collect medical information about your pregnancy and the birth and health of your baby. We want to follow you and your baby during the pregnancy and until delivery to try to learn if the study treatment has any effect on your pregnancy. We would like to follow the health of your baby at least at 6 and 12 months of age for any important medical issues.

#### What are the possible risks of staying in the study?

Your study doctor will explain the risks of the treatment for yourself, your pregnancy, your fetus and/or your future baby. You will be given a paper (leaflet) that summarizes the main side effects when used during pregnancy.

All the other risks (side effects) were explained to you when taking your consent for participation in the study.

Your privacy will be protected as detailed in the research consent form you have already signed.

## Are there benefits to staying in the study?

If your study doctor proposes that you stay in the study, s/he believes that the possible benefits of staying in the study and receiving the study treatment are bigger than the risks for you and your baby.

You will receive more treatment support in the study than you would outside the study and your pregnancy will be closely monitored.

Others with MDR-TB may benefit in the future from what we learn in this study. We hope that the information we gather about your pregnancy while taking the study drugs and after will help future patients and their children by increasing what we know about the possible of the study medicines on pregnant women and developing babies.

#### What should I do if I want to stop being in the study?

If you decide to stop being in the study, we will make sure you stop the study safely.

We will talk to you about follow-up care you might need, and you will be to come back at least for one additional study visit.

## **Treatment during pregnancy Consent Form**

Version 4.3 Version Date: 05 Jul 2022

SUBJECT IDENTIFICATION

And, we will tell you if we learn any new information that could make you change your mind and choose to leave the study.

If you decide to stop participating in the study, the study doctor will ask you for permission to collect information about your pregnancy and its outcome, and the condition of your newborn (at least at 6 and 12 months of age for any important medical issues).

Information collected from you will be used to help answer study questions. When you leave the study, your information may still be used for the study. If you do not want this information to be used, and you want it to be destroyed, please contact your study doctor or the email address endTB.clinicaltrial@paris.msf.org.

Also, your study doctor, at any point in time after your consent, might ask you to leave the study before you finish it. This may happen for example if s/he thinks that the risks of staying in the study are becoming higher than the expected benefits, or if s/he thinks that you need to receive treatment not allowed by the research study. If this happens, your study doctor will explain in detail all the reasons for his/her decision.

### Will I be paid or have to pay additional expenses if I stay in this research study?

You will not receive reimbursements in addition to the ones you already receive for taking part into the study. This study will not cover any costs from your pregnancy, delivery or care of your baby [to be adapted locally]. There will be no cost [or payment] to you if you stay in the study.

# What happens if my baby is injured or I am injured as a result of taking part in this research study?

If you or your baby suffer injury directly as a result of participation in this study, the sponsor has made insurance arrangements to pay for any injury you may suffer [or any miscarriage or damage to the fetus or your baby].

If this happens, please tell your study doctor and seek medical attention right away. The sponsor will ensure that you receive appropriate medical treatment for it and that your pregnancy course is closely monitored.

In an emergency, the sponsor has made plans to pay for a specialist, visit, related treatment, and/or a hospital stay. For non-urgent situations, the sponsor might pay for your visit to see a specialist. The study team will review your situation and decide whether the sponsor will pay for the resulting treatment if your condition is not the result of your participation in the study. You do not waive any of your legal rights by signing this consent form.

#### Who can I speak to if I have questions, concerns or complaints?

If you have questions about this study, you can contact [PI Name and title] at [PI telephone number]. You can also call [Clinical Investigator] at [CI number] with questions about this research study. If you have questions about the scheduling of appointments, call [Study Coordinator] at [SC number].

If you want to speak with someone not directly involved in this research study, please contact the [*Research Center IRB*] office. You can call them at [*Research Center IRB number*].

# **Treatment during pregnancy Consent Form**

Version 4.3 Version Date: 05 Jul 2022 SUBJECT IDENTIFICATION

#### **Informed Consent and Authorization**

Your signature on this document means the following:

I have read this consent form. It has been explained to me why I'm being asked to sign this informed consent, the risks and the possible benefits for the fetus and for me resulting from staying in the study. I have had the opportunity to ask questions. I understand the information given to me. I recognize that my participation is voluntary and that I can refuse or end my participation at any time, without any loss of benefits that I would otherwise have. I recognize that by signing this document, I do not lose any of my legal rights as a patient.

I will receive a complete, signed, dated copy of this informed consent form.

| I will receive a complete, signed, dated copy of th | is informed consent form. | |
|---|---|---|
| By signing below, I freely agree to continue my to take the study treatment that will be prescribed | <u> </u> | and I agree |
| Signature or thumbprint of pregnant participant | Date (DD/MMM/YYYY) | Γime |
| Name of pregnant participant, printed in capital le | itters | |
| If applicable, Signature of witness | Date (DD/MMM/YYYY) | Time |
| Name of witness, printed in capital letters | | |
| Study representative who obtained informed co | onsent: | |
| I have explained to the pregnant participant participate in the study and the risks for herself a have answered all of her questions. She understand accepts voluntarily to keep participating in the | nd the fetus deriving from the drug<br>nds the information described in the | gs intake and |
| Signature of representative | Date (DD/MMM/YYYY) | Time |
| Name of study representative, printed in capital le | etters | |
| 1 of stady representative, printed in cupital re | | |